CLINICAL TRIAL: NCT02920424
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of JNJ-56022473 in Subjects With Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of JNJ-56022473 in Subjects With Systemic Lupus Erythematosus
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision is based on a change in the benefit risk assessment of this drug for the lupus population targeted in this study.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108216; 2016-001260-11 (EudraCT Number); 56022473SLE1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: JNJ-56022473 or Placebo (4:1) (Experimental): Subjects will receive 3 subcutaneous (SC) administrations of the same dose level of JNJ-56022473 Dose 1, Dose 2, or Dose 3 or placebo every 2 weeks (in the ratio of 4:1 [4 active: 1 placebo]).
  Interventions: Drug: JNJ-56022473; Drug: Placebo
- Part B: JNJ-56022473 or Placebo (5:1) (Experimental): Subjects will receive 3 SC administrations of the same dose level of JNJ-56022473 or placebo every 2 weeks (in the ratio of 5:1 [5 active: 1 placebo]). The dose level(s) will be based upon an interim analysis (IA) of the Part A data.
  Interventions: Drug: JNJ-56022473; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-56022473 — Subjects will be administered with JNJ-56022473 SC depending upon on the dose levels.
Drug: Placebo — Subjects will receive matching placebo.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of JNJ-56022473 following multiple subcutaneous (SC) study agent administrations in subjects with Systemic Lupus Erythematosus (SLE) and to determine whether premedication with corticosteroids is required to improve the tolerability of SC JNJ-56022473.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a body weight in the range of 40 to 100 kilogram (kg), inclusive, and have a body mass index (BMI) of 18 to 32 kilogram per meter square (kg/m^2), inclusive, at screening
* Subjects eligible for enrollment in this study must qualify as follows: a) must meet Systemic Lupus International Collaborating Clinics (SLICC) criteria for diagnosis of lupus and b) must have at least one non-serologic clinical activity defined by the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) within 3 months prior to first study agent administration
* Have a positive gene signature score during screening, prior to first administration of study agent
* Subjects using allowed pre-existing lupus treatments, if stable for at least 6 weeks prior to the first dose of study medication:

  1. oral corticosteroids equivalent to an average dose up to or equal to (<=) 10 milligram (mg) of prednisone/day
  2. use of antimalarials (such as chloroquine or hydroxychloroguine) for at least 8 weeks
  3. maximum of 1 non-corticosteroid immunosuppressive drug

Exclusion Criteria:

* Subject with history or suspected occurrence of drug-induced systemic lupus erythematosus (SLE)
* Subject has unstable lupus nephritis and/ or has active Central nervous system (CNS) lupus or history of severe CNS lupus, including but not limited to seizures, psychosis, transverse myelitis, CNS vasculitis and optic neuritis
* Major surgery prior to, and, if planned, during and shortly after the study is not eligible
* Subject has or has had an acute illness, including a common cold, within 2 weeks prior to the study agent administration or has had a major illness or hospitalization within 4 months prior to the screening visit
* Any other inflammatory diseases that might confound the evaluations of efficacy are excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-30 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-09-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects With Treatment-Emergent Adverse Events (TEAEs) by Severity and Serious Adverse Events (SAEs) Through Week 16 | Up to 16 weeks
Percentage of Subjects With Grade 1, Grade 2, and Grade 3 Systemic Administration-Related Reactions (SARR) After Drug Administration | Up to 16 weeks

SECONDARY OUTCOMES:
Serum Concentration of JNJ-56022473 | Up to 16 weeks
Number of Subjects With Presence of Anti-JNJ-56022473 Antibodies | Up to 16 weeks
Gene Expression Measured in Whole Blood by Quantitative Polymerase Chain Reaction (qPCR) | Up to 38 weeks
  Whole blood samples collected from subjects enrolled in this study will be examined by qPCR to assess the ability of JNJ-56022473 to initiate the expected effect on target cells.
Counts of Target Cells | Up to 38 weeks
  Counts of target cells will be measured by flow cytometry from whole blood.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- Germany (3):
  - Charité Research Organisation GmbH, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz